CLINICAL TRIAL: NCT05352204
Title: The Guiding Value of Tumor Micronecrosis for Using Postoperative Transcatheter Arterial Chemoembolization in Patients With Hepatocellular Carcinomas
Brief Title: Effect of Tumor Micronecrosis on Postoperative Transcatheter Arterial Chemoembolization in Patients With Hepatocellular Carcinomas
Status: Completed | Type: Observational
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, TingBo Liang, FACS, Zhejiang University
Other Study IDs: PTHCC
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Carcinoma, Hepatocellular
Keywords: hepatocellular carcinoma; TACE; tumor necrosis
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- micronecrosis(+) group
  Interventions: Procedure: transcatheter arterial chemoembolization
- micronecrosis(-) group

INTERVENTIONS:
Procedure: transcatheter arterial chemoembolization — transcatheter arterial chemoembolization after liver resection
  Groups: micronecrosis(+) group

SUMMARY:
Micronecrosis is a novel pathological feature of hepatocellular carcinoma (HCC). This study was aimed at evaluating the effect of tumor micronecrosis on postoperative transcatheter arterial chemoembolization (TACE) in patients with hepatocellular carcinomas, and further exploring the value of micronecrosis for guiding TACE in HCC management.

ELIGIBILITY:
Inclusion Criteria:

* (1) pathologically confirmed HCC (2) achievement of R0 resection.

Exclusion Criteria:

* (1) simultaneous presence of other tumors ; (2) receipt of preoperative anti-tumoral treatments; (3) concurrent treatment with other antitumoral therapies in combination with TACE; (4) tumor necrosis that could be observed by gross examination; (5) a lack of necessary preoperative laboratory test results.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: From June 2014 to April 2018, HCC patients who underwent liver resection in our center were retrospectively reviewed.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Actual)
Dates: Start 2020-04-30 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-04-14 (Actual)

PRIMARY OUTCOMES:
overall survival | after liver resection until June 1, 2020
  the number of months from the date of surgery to the date of the last follow-up visit or time of death.

SECONDARY OUTCOMES:
disease-free survival | after liver resection until June 1, 2020
  the number of months from the date of surgery to the date of first confirmable recurrence or death

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - the First Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - the First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang